CLINICAL TRIAL: NCT01553474
Title: Blood and Saliva Sample Collection and Submission to the Age-Related Eye Disease Study 2 (AREDS2) Genetic Repository
Brief Title: Blood and Saliva Sample Collection for AREDS 2
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120085; 12-EI-0085
Record Dates: First submitted 2012-03-13; First posted 2012-03-14 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2013-02-05

CONDITIONS: Age-Related Macular Degeneration; Eye Diseases
Keywords: Age-Related Macular Degeneration (AMD); Eye Diseases
MeSH Terms: conditions — Macular Degeneration; Eye Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The Age-Related Eye Disease Study 2 (AREDS 2) is looking at different eye diseases. Study participants will provide blood and saliva samples. The samples will be stored for research on eye diseases.

Objectives:

- To collect blood and saliva samples for AREDS 2 research.

Eligibility:

- AREDS 2 research study participants.

Design:

* Participants will provide blood and saliva samples.
* The samples will be submitted with personal and medical information. This information will be collected during the AREDS 2 procedures.

DETAILED DESCRIPTION:
AREDS2 is a multi-center, Phase III, randomized clinical trial designed to assess the effects of oral supplementation of high doses of macular xanthophylls (lutein and zeaxanthin) and/or omega-3 long-chain polyunsaturated fatty acids (LCPUFAs) as a treatment for age-related macular degeneration (AMD), cataract and moderate vision loss. In addition to this objective, the AREDS2 study will provide information on the clinical course, prognosis, and risk factors for development and progression of both AMD and cataract. Other study goals include the evaluation of eliminating beta-carotene and/or reducing zinc in the original AREDS formulation on the progression and development of AMD. AREDS2 will also seek to validate the fundus photographic AMD scale developed from AREDS.

The objective of this protocol is to have AREDS2 participants submit blood and saliva samples to the AREDS2 Genetic Repository (Fisher BioServices, Rockville, MD) in order to provide further materials for the study of the genetic and biochemical bases for eye disease and possibly other diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they were enrolled in the AREDS2 protocol and willing to have their blood drawn and saliva collected.

EXCLUSION CRITERIA:

Participants will not be eligible if they were not enrolled in AREDS2 and are not willing to have their blood drawn and saliva collected.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-02-24; Study Completion 2013-02-05

CONTACTS AND LOCATIONS:
Overall Officials: Wai T Wong, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States